CLINICAL TRIAL: NCT01393314
Title: A Randomized Controlled Trial of Telemonitoring in Older Adults With Heart Failure
Brief Title: A Trial of Telemonitoring in Adults With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1KL2RR024990 - 2; 1KL2RR024990 (NIH)
Record Dates: First submitted 2011-07-01; First posted 2011-07-13 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Honeywell HomMed Telemonitor (Active Comparator): TeleCareOhio Monitor (Honeywell HomeMed) system provides in-home medical monitoring for patients with chronic disease such as heart failure.
  Interventions: Device: Honeywell HomMed Telemonitor
- Usual care (No Intervention): These participants receive usual care which consists of usual home-care with educational package.

INTERVENTIONS:
Device: Honeywell HomMed Telemonitor — telemonitoring post hospitalization
  Arms: Honeywell HomMed Telemonitor

SUMMARY:
This is a randomized controlled trial of telemonitoring vs usual care provided by home care agencies for patients with heart failure.

The study hypothesis is that Telemonitoring will reduce hospital re-admission rates, urgent care visits, unscheduled physician appointments, Emergency Room visits in patients with heart failure over the 60 day post hospitalization period.

DETAILED DESCRIPTION:
A 60 day stratified, randomized clinical trial of a home-based telemonitoring system (TEP) vs. usual home-care with educational package (EP). Both Groups will receive intensive patient education and primary care physicians will be prompted to adhere to heart failure management guidelines. The study will be conducted on 100 patients receiving home care nursing services post-hospital discharge.

Each participant will be randomized in equal amounts to treatment (TEP) or no treatment (EP).

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure (primary or secondary) diagnosis regardless of ejection fraction (EF) and New York Heart Association (NYHA) class II- IV at the time of Home Health Care (HHC) admission and HHC services initiated following a hospital stay

Exclusion Criteria:

* Inability to stand on a scale, weight over 500 pounds, unable to hear and/or see, or no working land line phone in the residence.
* Additional exclusion criteria were: patients with severe ischemic heart disease, Myocardial Infarction (MI) and/or Coronary artery bypass graft surgery(CABG) in the last 6 weeks, severe uncorrected valvular disease, home inotropic therapy, severe lung disease (oxygen dependent), active cancer, uncorrected thyroid disease, AIDS, or end stage renal disease on dialysis.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Boxer, MD, Principal Investigator — Case Western Reserve Univeristy

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care which consists of usual home-care with educational package.
Period: Overall Study
Arm/Group | Honeywell HomMed Telemonitor | Usual Care
Started | 54 | 45
Completed | 54 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Honeywell HomMed Telemonitor: TeleCareOhio Monitor (Honeywell HomeMed) system provides in-home medical monitoring for patients with chronic disease such as heart failure; telemonitoring post hospitalization.
- Total: Total of all reporting groups
Arm/Group | Honeywell HomMed Telemonitor | Usual Care | Total
Number analyzed (Participants) | 54 | 45 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (12.1) | 74.7 (11.3) | 74.85 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 27 | 67
  Male | 14 | 18 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 45 | 33 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Time Participants Are Readmitted to the Hospital or Visit the Emergency Department (ED).
Description: Median time to combined endpoint to see if/when the participants need to be readmitted to the hospital or visit the ED
Time Frame: Participants were followed for the duration of home care services up to 12 months
Measure: Median (Standard Deviation); unit: Days
Groups:
- Usual Care: This participants receive usual care which consists of usual home-care with educational package.
Arm/Group | Honeywell HomMed Telemonitor | Usual Care
Number analyzed (Participants) | 54 | 45
Days | 60 (3) | 62 (8.5)

2. Secondary Outcome: Kansas City Cardiomyopathy Questionaire
Description: Health Status, Change in Overall Summary Score minimum: 0 maximum: 100 higher scores=better outcome
Time Frame: Participants were followed for the duration of home care services up to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Honeywell HomMed Telemonitor | Usual Care
Number analyzed (Participants) | 54 | 45
score on a scale | 34.3 (12.9) | 28.3 (16.85)

ADVERSE EVENTS:
Arm/Group | Honeywell HomMed Telemonitor | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/45
Other Adverse Events (participants affected / at risk) | 0/54 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No